CLINICAL TRIAL: NCT06797180
Title: Effectiveness of Virtual Reality-Based Educational Intervention in Enhancing Caregiving Competence for Managing Agitated Behaviors in Dementia Residents: A Randomized Controlled Trial
Brief Title: VR-Based Intervention for Caregiving Competence in Dementia
Acronym: VRE-ABC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MMC-RD-112-1B-P004; MOST 111-2314-B-715-004-MY3 (Other Grant/Funding Number: National Science and Technology council)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Competence
Keywords: Behavioral and Psychological Symptoms of Dementia (BPSD); Caregiving Competence; Dementia Care; Virtual Reality Education; Residential care homes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- This group will receive BPSD foundational education followed by VR-based training. (Experimental): The intervention consists of two components:
  1. BPSD Foundational Education: A 100-minute educational session covering an overview of BPSD, identification of common symptoms, strategies for managing BPSD, and the role of caregivers.
  2. VR-based Training: A 100-minute VR-based training, including 20 minutes of immersive VR scenarios to experience at least two types of BPSD, 20 minutes of group discussion to share practical strategies, and 20 minutes of evidence-based explanation of management techniques, 15 minutes for scenario reflection, and 25 minutes for Q&A and summarization.
  Interventions: Device: Virtual Reality Education for Dementia Caregivers
- This group will only receive BPSD foundational education. (No Intervention): The control group will only receive the 100-minute BPSD foundational education, which covers the same topics as the experimental group but without the VR-based training.

INTERVENTIONS:
Device: Virtual Reality Education for Dementia Caregivers — This group will receive 100 minutes of BPSD foundational education followed by 100 minutes of VR-based training focused on managing BPSD.
  Arms: This group will receive BPSD foundational education followed by VR-based training.

SUMMARY:
This study aims to develop and evaluate the effectiveness of a VR-based educational intervention designed to improve the dementia caregiving abilities of formal caregivers in residential care homes. The intervention focuses on enhancing caregivers' knowledge and skills in managing behavioral symptoms of dementia through immersive VR scenarios, group discussions, and evidence-based management strategies, with the goal of better equipping them to provide high-quality care for residents with dementia.

DETAILED DESCRIPTION:
Background:

Agitated behaviors, such as aggression, care resistance, and wandering, are common in dementia and present significant challenges for formal caregivers in long-term care (LTC) facilities. These behaviors often stem from unmet needs, such as pain, discomfort, or communication barriers, contributing to caregiver stress and reduced care quality. Virtual reality (VR) technology offers an immersive, first-person experience that enables caregivers to better understand triggers of agitated behaviors, empathize with residents' experiences, and improve their caregiving abilities.

Purpose:

This study aims to develop and evaluate the effectiveness of a VR-based educational intervention for formal caregivers in residential care homes. Specifically, the study compares two groups: (1) an experimental group receiving both a 100-minute behavioral and psychological symptom (BPSD) foundational education and an additional 100-minute VR training program, and (2) a control group receiving only the 100-minute BPSD foundational education. The study evaluates three outcomes: (1) dementia care competence, (2) confidence in caregiving, and (3) self-reported frequency of BPSD assessment and management at pre-intervention, post-intervention, and two-week follow-up.

Methods:

The VR scenarios and training intervention were developed through a systematic literature review, four focus group interviews with formal caregivers, and pilot testing in a residential LTC facility in Northern Taiwan. A single-blind randomized controlled trial with repeated measures design was conducted across six LTC facilities. The experimental group received 100 minutes of BPSD foundational education, covering an overview of BPSD, identification of common symptoms, strategies for managing BPSD, and the role of caregivers. Additionally, they participated in 100 minutes of VR-based training, which included 20 minutes of immersive VR scenarios to experience at least two types of BPSD, 20 minutes of group discussion to share practical strategies, 20 minutes of evidence-based explanation of management techniques, 15 minutes for scenario reflection, and 25 minutes for Q&A and summarization. The control group, however, only received the 100-minute BPSD foundational education without the VR component. Resident data, including demographics, medical conditions, and Barthel Index scores, were collected. Outcome measures included the Dementia Competence Scale (DCS) , self-reported confidence in caregiving and weekly self-reported BPSD assessment and management frequencies. Data analysis utilized SPSS 25.0, applying descriptive statistics and mixed linear models to examine within- and between-group improvements over time.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Able to communicate in Mandarin or Taiwanese.
3. A formal caregiver of individuals with dementia.
4. At least one month of work experience in the residential care facility.

Exclusion Criteria:

1. Caregivers who do not meet the above inclusion criteria.
2. Individuals who are unable or unwilling to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in caregiving ability scores before intervention to post-intervention and follow-up. | Data will be collected before the intervention (baseline), immediately post-intervention (after training), and at follow-up (two weeks after the intervention).
  Caregiving ability was measured using the Dementia Competence Scale for Acute Care (DCS) developed by Yang, Yang, Hsiao, Kuo, and Wang (2021). This scale includes three subscales: 13 items on knowledge, 11 items on attitudes, and 9 items on skills. The Cronbach's α values for the knowledge, attitude, and skills subscales were 0.88, 0.94, and 0.85, respectively. The test-retest reliability, as measured by the intraclass correlation coefficient (ICC), was 0.82 for the overall scale, with 0.87 for the knowledge subscale, 0.64 for the attitude subscale, and 0.74 for the skills subscale.
Confidence in assessing and managing BPSD | Data will be collected before the intervention (baseline), immediately post-intervention (after training), and at follow-up (two weeks after the intervention).
  Confidence in assessing BPSD (Behavioral and Psychological Symptoms of Dementia) and in effectively managing BPSD was evaluated using a 5-point scale, ranging from "very unconfident" to "very confident."

SECONDARY OUTCOMES:
Change in frequency of assessment and management of BPSD before intervention to post-intervention and follow-up. | Data will be collected before the intervention (baseline), at 1 week post-intervention, and at follow-up (two weeks after the intervention).
  This measure includes the frequency of:
  Assessment and documentation of dementia-related problem behaviors over the past week.
  Pharmacological interventions, non-pharmacological interventions, and the referral frequency for dementia-related behaviors over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — School of Nursing
Locations (1):
- Department of Nursing, New Taipei City, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No